CLINICAL TRIAL: NCT02526914
Title: Effects of Intranasal Oxytocin and Vasopressin on Social Behavior and Decision Making
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: David Mankuta (Other)
Collaborators: Hebrew University of Jerusalem (Other)
Responsible Party: Sponsor-Investigator, David Mankuta, David Mankuta, MD, Hadassah Medical Organization
Organization: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Hadassah Medical Organization
Record Dates: First submitted 2015-08-14; First posted 2015-08-18 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-08

CONDITIONS: Healthy
Keywords: social cognition; oxytocin; vasopressin; decision making; social decision making; economic games
MeSH Terms: conditions — Diabetes Insipidus | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intranasal Oxytocin (Experimental): Participants will self-administer 24 IU Oxytocin. 5 puffs per nostril (1 puff = 2.5 IU Oxytocin).
  Interventions: Drug: Intranasal Oxytocin
- Intranasal vasopressin (Experimental): Participants will self-administer 20 IU vasopressin. 5 puffs per nostril (1 puff = 2 IU vasopressin).
  Interventions: Drug: Intranasal vasopressin
- Intranasal placebo (Placebo Comparator): contains all the ingredients as in the oxytocin and vasopressin conditions, save for the active ingredient. Participants will self-administer 5 puffs per nostril.
  Interventions: Drug: Intranasal placebo

INTERVENTIONS:
Drug: Intranasal Oxytocin — Through the use of 2ml bottles attached with metered nasal pumps (1 puff = .1ml), participants will self-administer 24 IU Oxytocin. 5 puffs per nostril (1 puff = 2.5 IU Oxytocin).
  Other Names: syntocinon
  Arms: Intranasal Oxytocin
Drug: Intranasal vasopressin — Through the use of 2ml bottles attached with metered nasal pumps (1 puff = .1ml), participants will self-administer 20 IU vasopressin. 5 puffs per nostril (1 puff = 2 IU vasopressin).
  Arms: Intranasal vasopressin
Drug: Intranasal placebo — Through the use of 2ml bottles attached with metered nasal pumps (1 puff = .1ml), participants will self-administer 5 puffs per nostril. Placebo consists of: di-sodium hydrogen phosphate, critic acid, sodium chloride, glycerin, benzalkonium chloride and aqua bidest.
  Arms: Intranasal placebo

SUMMARY:
The purpose of this study is to investigate the role of a one-time intranasal administration of the oxytocin, vasopressin, or placebo on prosocial decision making such as cooperation and competition in a healthy population of student controls.

ELIGIBILITY:
Inclusion Criteria:

• healthy controls

Exclusion Criteria:

* Past or present psychiatric, neurological, endocrinological or severe chronic medical illness.
* Use of medications or drugs that would interfere with study results. This includes steroids, medications for psychiatric symptoms like anxiety or depression, stimulants, and medications for high blood pressure. Participants will be asked to tell the investigators of any medications or drugs that they are taking. The investigators will consider the drug interactions with oxytocin and vasopressin prior to study, and participants will not be able to participate in the study if the drug interactions could be dangerous.
* history of drug or alcohol addiction
* Pregnancy or Nursing Status: Because of the risk to an unborn fetus or infant, women who are pregnant or nursing are excluded from this protocol. All females will have a pregnancy test performed no more than 24 hours before each drug administration and will not be able to participate if the pregnancy test is positive.

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 432 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-07 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Preferences for competitive vs cooperative compensations and monetary allocations as measured by participants monetary allocations and compensation choice | approximately 45 minutes after intranasal administration of vasopressin, oxytocin, or placebo
  A group analysis will compare compensations preference (competitive vs. noncompetitive), performance and outcomes and monetary allocations on several economic games between the oxytocin, vasopressin and placebo groups.

SECONDARY OUTCOMES:
Redistribution preferences as measured by participants' tax rate determination | approximately 45 minutes after intranasal administration of vasopressin, oxytocin, or placebo
  Participants will choose redistribution of monetary units by determined tax rate (high vs. low). Each participant gets a different amount of monetary units (ranging from 10 to 150). Using a mixed 2 (above vs. below group mean of monetary units) x 3 (oxytocin, vasopressin, placebo) factorial design, comparisons of these tax rate preference will then be made for those in the oxytocin vs. vasopressin vs. placebo groups. Main effects of drug condition (oxytocin, vasopressin, placebo) and monetary condition (above, below group mean), as well as an interaction between drug condition and monetary condition will be analyzed at a significance level of p<.05.
Willingness to compete as measured by participants compensation choice. | approximately 45 minutes after intranasal administration of vasopressin, oxytocin, or placebo
  Willingness to compete will be measured by participants' preference whether to compete against other participant for a monetary payment or to get a smaller payment for their non-competitive piece rate performance on maze solving task. We will analyses performance and payment preference (competitive vs. noncompetitive) between oxytocin, vasopressin and placebo at a significance level of p<.05.
Monetary offers in public goods game | approximately 45 minutes after intranasal administration of vasopressin, oxytocin, or placebo
  Participants in two rival teams will offer monetary units for the right to take part in a lottery (higher team's offer = higher odds to win). Members of each team may, for a monetary cost, impose a tax on their team members. We will compare monetary offers and taxes' impose pattern between oxytocin, vasopressin and placebo groups at a significance level of p<.05 .
Bargaining performance as assessed by participants' earnings in bargaining compensation | approximately 45 minutes after intranasal administration of vasopressin, oxytocin, or placebo
  Analysis will compare negotiation outcomes, in terms of monetary units earnings between oxytocin, vasopressin and placebo groups at a significance level of p<.05.
Monetary offers in all pay auction | approximately 45 minutes after intranasal administration of vasopressin, oxytocin, or placebo
  Analysis will compare participants' monetary offers in multi-participants all-pay auction between oxytocin, vasopressin and placebo groups at a significance level of p<.05.
Negative hypothesis test strategy usage on Wason's-rule-discovery-task after exposure to trustworthy/untrustworthy face | approximately 45 minutes after intranasal administration of vasopressin, oxytocin, or placebo
  Number of positive hypothesis tests (compare to 'negative-test') out of 6 participants' generated tests. Analysis will compare number of positive tests (vs. negative tests) between oxytocin, vasopressin and placebo groups at a significance level of p<.05.
Positive and negative affect scale (PANAS) | approximately one hour and fifteen minutes after administration of oxytocin, vasopressin or placebo
  Using the Positive and negative affect scale (PANAS) we will measure participants emotional reaction to Oxytocin, vasopressin and placebo. Participants will report their current mood by rate the level they feel 20 different emotions at the moment on a the PANAS scale, ranging from 1 (not at all) to 5 (very much).
Fear of negative evaluation (FNE) as measured by self reporting | approximately one hour and fifteen minutes after administration of oxytocin, vasopressin or placebo
  Participants will report their fear of evaluation by rate how much 12 statements characterize them. participants will use a scale ranging from 1 ("Not at all characteristic me") to 5 ("Extremely characteristic of me").
Social value orientation as measured by monetary allocations preferences | approximately one hour and fifteen minutes after administration of oxytocin, vasopressin or placebo
  Participants will make decisions regarding the allocation of monetary units between themselves and other participants. We will measure the quantity of monetary units kept for themselves vs. given to other participants.

CONTACTS AND LOCATIONS:
Overall Officials: David Mankuta, MD, Principal Investigator — Hadassah University Medical Organization
Locations (1):
- Hadassah University Medical Organization, Jerusalem, Jerusalem, Israel

REFERENCES:
- [Background] Meyer-Lindenberg A, Domes G, Kirsch P, Heinrichs M. Oxytocin and vasopressin in the human brain: social neuropeptides for translational medicine. Nat Rev Neurosci. 2011 Aug 19;12(9):524-38. doi: 10.1038/nrn3044. PMID 21852800
- [Background] Kosfeld M, Heinrichs M, Zak PJ, Fischbacher U, Fehr E. Oxytocin increases trust in humans. Nature. 2005 Jun 2;435(7042):673-6. doi: 10.1038/nature03701. PMID 15931222
- [Background] Veening JG, Olivier B. Intranasal administration of oxytocin: behavioral and clinical effects, a review. Neurosci Biobehav Rev. 2013 Sep;37(8):1445-65. doi: 10.1016/j.neubiorev.2013.04.012. Epub 2013 May 4. PMID 23648680